CLINICAL TRIAL: NCT07074249
Title: Anatomical Accuracy of Blind Dry Needling Procedures on the Lumbar Paraspinal Muscles: An Ultrasonography-Assisted Observational Study
Brief Title: Blind Needling Accuracy in Lumbar Muscles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, nurmuhammet tas, dr., Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: erzurum rtrh3
Record Dates: First submitted 2025-06-23; First posted 2025-07-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dry Needling Lumbar Paraspinal Muscles
Keywords: dry needling; ultrasound guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blind Dry Needling Lumbar Paraspinal Muscles (Experimental): All interventions will be performed by a physical medicine and rehabilitation specialist with clinical experience.
  * Targeted muscles:
  * *Iliocostalis lumborum (ICL)*
  * *Longissimus thoracis (LT)*
  * *Multifidus (M)*
  * Interventions will be performed from the right side, between the L2-L5 levels.
  * A total of *three different dry needling applications* will be performed for these three muscles for each participant.
  Interventions: Procedure: "Anatomical Accuracy of Blind Dry Needling Procedures on the Lumbar Paraspinal Muscles: An Ultrasonography-Assisted Observational Study"
- Ultrasound-Guided Needle Location Verification (Experimental): All interventions will be performed by a physical medicine and rehabilitation specialist with clinical experience. * Targeted muscles: * *Iliocostalis lumborum (ICL)* * *Longissimus thoracis (LT)* * *Multifidus (M)* * Interventions will be performed from the right side, between the L2-L5 levels. * A total of *three different dry needling applications* will be performed for these three muscles for each participant. After the needling procedure, a second clinician evaluates the needle's location in the muscle using ultrasonography.
  Interventions: Procedure: "Anatomical Accuracy of Blind Dry Needling Procedures on the Lumbar Paraspinal Muscles: An Ultrasonography-Assisted Observational Study"

INTERVENTIONS:
Procedure: "Anatomical Accuracy of Blind Dry Needling Procedures on the Lumbar Paraspinal Muscles: An Ultrasonography-Assisted Observational Study" — * All interventions will be performed by a physical medicine and rehabilitation specialist with clinical experience.
  * Targeted muscles:
  * *Iliocostalis lumborum (ICL)*
  * *Longissimus thoracis (LT)*
  * *Multifidus (M)*
  * Interventions will be performed from the right side, between the L2-L5 levels.
  * A total of *three different dry needling applications* will be performed for these three muscles for each participant.
Procedure: "Anatomical Accuracy of Blind Dry Needling Procedures on the Lumbar Paraspinal Muscles: An Ultrasonography-Assisted Observational Study" — *All interventions will be performed by a physical medicine and rehabilitation specialist with clinical experience. * Targeted muscles: * *Iliocostalis lumborum (ICL)* * *Longissimus thoracis (LT)* * *Multifidus (M)* * Interventions will be performed from the right side, between the L2-L5 levels. * A total of *three different dry needling applications* will be performed for these three muscles for each participant. After each intervention, the needle tip position will be evaluated by a second specialist with *high-resolution linear probe ultrasound*.

SUMMARY:
The aim of this study is to evaluate the accuracy of blinded invasive interventions (dry needling) on the deep paraspinal muscles of the lumbar region (iliocostalis lumborum, longissimus thoracis, and multifidus) to reach the anatomical target. The accuracy of the interventions will be evaluated observationally with ultrasonography after the procedure.

DETAILED DESCRIPTION:
*Method:*

* All interventions will be performed by a physical medicine and rehabilitation specialist with clinical experience.
* After each intervention, the needle tip position will be evaluated by a second specialist with *high-resolution linear probe ultrasound*.
* Targeted muscles:
* *Iliocostalis lumborum (ICL)*
* *Longissimus thoracis (LT)*
* *Multifidus (M)*
* Interventions will be performed from the right side, between the L2-L5 levels.
* A total of *three different dry needling applications* will be performed for these three muscles for each participant.
* When a total of *20 participants* is planned, *60 injection attempts* will be analyzed.
* Will be used only for post-hoc observational validation purposes.
* No pharmacological agent will be administered during the intervention, only dry needling will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65

  * Individuals with nonspecific low back or back pain and planned physical therapy
  * Individuals with suspected MPS, especially in the paraspinal muscles
  * Individuals with indications for dry needling
  * Those who can cooperate with the procedure and give written consent

Exclusion Criteria:

* * Anticoagulant use

  * History of spine surgery, deformity, severe scoliosis
  * Regional skin lesion or infection
  * Patients who cannot cooperate
  * Pregnancy
  * Serious systemic diseases such as malignancy or neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
"Anatomical Accuracy of Blind Dry Needling Procedures on the Lumbar Paraspinal Muscles: An Ultrasonography-Assisted Observational Study" | 2 week
  Correct placement rates will be calculated for each muscle. The agreement between the ultrasound and verification results of the blinded applications will be evaluated with Kappa statistics. Chi-square test or McNemar test will be used for differences between muscles.